CLINICAL TRIAL: NCT01172119
Title: A Prospective, Single Blinded, Randomized Study to Evaluate the Safety and Effictiveness of a Low and Standard Dose Biolimus A9TM Drug-Eluteing Coronary Stent Delivery System Compared With a TaxusTM LiberteTM Control Arm for Treatment of Stenotic Lesions in Native Coronary Arteries.
Brief Title: BioFreedom FIM Clinical Trial.
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Biosensors Europe SA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 08EU01
Record Dates: First submitted 2010-07-28; First posted 2010-07-29 (Estimated); Last update posted 2014-09-09 (Estimated); Status verified 2014-09

CONDITIONS: Treatment Of Stenotic Lesions In Native Coronary Arteries.
Keywords: Coronary Disease, Coronary Stenosis, Angioplasty, Coronary restenosis, Drug Eluting Stent
MeSH Terms: conditions — Coronary Disease; Coronary Stenosis; Coronary Restenosis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- BioFreedom Standard Dose (Experimental)
  Interventions: Device: Biofreedom Drug Eluting Stent
- BioFreedom Low Dose (Experimental)
  Interventions: Device: Biofreedom Drug Eluting Stent
- Taxus Liberte drug eluting stents (Active Comparator)
  Interventions: Device: Tuxus Liberte Drug Eluting Stent

INTERVENTIONS:
Device: Biofreedom Drug Eluting Stent — Biofreedom DES with a standard dose of Biolimus A9TM
  Arms: BioFreedom Standard Dose
Device: Biofreedom Drug Eluting Stent — Biofreedom DES with a low dose of Biolimus A9TM
  Arms: BioFreedom Low Dose
Device: Tuxus Liberte Drug Eluting Stent — Standard paclitaxel dose Taxus Liberte DES
  Arms: Taxus Liberte drug eluting stents

SUMMARY:
Prospective, multi center, randomized, single blinded study designed to demonstrate the safety and effectiveness of the Biosensors BioFreedom Drug-Eluting Coronary Stent Delivery System at multiple time points compared to the Taxus Liberte DES in the treatment of single de novo native coronary artery lesions ranging in diameter from ≥2.5 mm to ≤3.0 mm and ≤ 14 mm in length.

ELIGIBILITY:
Inclusion Criteria:

* The subject is >18 years of age.
* The subject is an acceptable candidate for PTCA, stenting, and emergent CABG.
* Patients with multiple lesions as long as the last lesion to be treated fits the Inclusion criteria of the target lesion.
* The subject must have clinical evidence of ischemic heart disease or a positive functional study.
* The study stent target vessel must be a native coronary artery with a stenosis of >50% and <100%.
* The study stent target vessel reference diameter must be >2.5 mm and ≤ 3.0 mm.(Measurements may be made by careful visual estimate or on-line quantitative coronary angiography.)
* The study stent target lesion is a de novo lesion that has not been previously stented.
* The study stent target lesion must be ≤ 14 mm in length thus allowing for adequate lesion coverage with a single stent.
* The subject is male or, if female, is either not of childbearing potential or has had a negative pregnancy test within seven (7) days prior to the procedure.
* The subject or the subject's legal representative has been informed of the nature of the study and has provided written informed consent as approved by the Institutional Ethics Committee (IEC) of the clinical site.
* The subject and the treating physician agree that the subject will return for all required post-procedure follow-up visits.

Exclusion Criteria:

* Multiple lesions to be treated in the same target vessel.
* Patients who require more than one BioFreedom stent except that an additional BioFreedom stent may be implanted in the target lesion for geographic miss or bailout
* A documented left ventricular ejection fraction < 30% assessed within 6 months prior to procedure by echocardiography, during a previous angiography or as measured during pre-procedure angiography.
* A known hypersensitivity or contraindication to aspirin, heparin, bivalirudin, ticlopidine and, clopidogrel, stainless steel, Biolimus A9, Paclitaxel or a sensitivity to contrast media, which cannot be adequately pre-medicated.
* A platelet count <100,000 cells/mm³ or >700,000 cells/mm³, or a WBC <3,000 cells/mm³.
* Evidence of an acute myocardial infarction within 72 hours of the intended treatment (defined as: Q wave or non-Q wave infarction having CK enzymes > 2 times the upper laboratory normal with the presence of a CK-MB elevated above the institutions upper limit of normal).
* A previous coronary interventional procedure was performed either a.) within 24 hours prior to the procedure or b.) within 12 months prior to the procedure for any lesion in the target vessel.
* The subject requires planned interventional treatment of any lesion in either the target vessel within 12 months or in any non-target vessel within 30 days post-procedure.
* The target and non-target lesion require treatment with a device other than PTCA prior to stent placement (such as, but not limited to, directional coronary atherectomy, excimer laser, rotational atherectomy, etc.).
* The target vessel has angiographic evidence of thrombus or is excessively (2 bends > 90º to reach the target lesion) tortuous.
* The target lesion has any of the following characteristics:

  1. Lesion location is aorto-ostial, left main coronary artery, or within 5 mm of the origin of the LAD, LCX, or RCA.
  2. Is at a >45º bend in the vessel.
  3. Is moderately to severely calcified (visible by fluoro).
* Stenting of the target or non-target lesion would "jail" or cover a side branch >2.0 mm in diameter or occur at the ostium of the sidebranch.
* History of a stroke or transient ischemic attack (TIA) within the prior 6 months or permanent neurologic deficit.
* History of upper GI bleeding within the prior 6 months.
* The subject has a history of bleeding diathesis or coagulopathy or will refuse blood transfusions.
* Concurrent medical condition with a life expectancy of less than 18 months.
* Currently participating in an investigational drug or another device study that has not completed the primary endpoint or that clinically interferes with the current study endpoints. [Note: Trials requiring extended follow-up for products that were investigational, but have since become commercially available, are not considered investigational trials.]
* Any contraindications as mentioned in the TaxusTM LiberteTM Instructions for Use (IFU).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 182 (Actual)
Dates: Start 2008-08; Primary Completion 2010-06 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
In-Stent Late Lumen Loss at 12 months post-procedure. | 12 Months

SECONDARY OUTCOMES:
In-Stent Late Lumen Loss (LL) at 4 months post-procedure for patients receiving IVUS/Angio at 4 months | 4 months
2. Major adverse cardiac events (MACE) at 30 days, defined as death, myocardial infarction or ischemic target vessel revascularization (PCI or CABG). | 30 days
3. Major Adverse Cardiac Event (MACE) at hospital discharge, 30 days, 4 months, 12 months, and 2, 3, 4 and 5 years post-procedure. | 5 years
Vascular complications through hospital discharge. | 5 years
5. Rates of stent thrombosis, per ARC definition of definite and probable and categorized as early, late or very late, at 30 days, 4 and 12 months, 2, 3, 4 and 5 years post-procedure. | 5 years
6. Biolimus A9 drug systemic drug levels post-procedure, 4 hours post-procedure, at hospital discharge, and at 30 days and 4 months clinical follow-up. | 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Eberhard Grube, Prof Dr med, Principal Investigator — Department of Cardiology Hospital Alemao O. Cruz, Sao Paulo, Brazil
Locations (4):
- Germany (4):
  - Medical Care Center, Hamburg University Cardiovascular Center, Hamburg
  - Herzzentrum Leipzig GmbH, Leipzig
  - HELIOS - Klinikum Siegburg, Siegburg
  - Krankenhaus der Barmherzigen Brüder, Trier

REFERENCES:
- [Derived] Costa RA, Abizaid A, Mehran R, Schofer J, Schuler GC, Hauptmann KE, Magalhaes MA, Parise H, Grube E; BioFreedom FIM Clinical Trial Investigators. Polymer-Free Biolimus A9-Coated Stents in the Treatment of De Novo Coronary Lesions: 4- and 12-Month Angiographic Follow-Up and Final 5-Year Clinical Outcomes of the Prospective, Multicenter BioFreedom FIM Clinical Trial. JACC Cardiovasc Interv. 2016 Jan 11;9(1):51-64. doi: 10.1016/j.jcin.2015.09.008. PMID 26762911